CLINICAL TRIAL: NCT06040918
Title: Single Center Study Evaluating The Effects Of N-803 Stimulation On The Expansion, Enrichment, And Proliferation Of Natural Killer Cells Collected By Apheresis
Brief Title: Single Center Study Of N-803 Stimulation On Expansion, Enrichment, Proliferation Of Natural Killer Cells Collected By Apheresis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: QUILT-105
Record Dates: First submitted 2023-06-26; First posted 2023-09-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — ALT-803

STUDY DESIGN:
Intervention Model Description: Up to 10 healthy subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Subjects (Experimental): Subjects will be scheduled for first apheresis collection on study Day 1. All subjects will receive N-803 at a fixed dose of 1 mg by subcutaneous (SC) injection 4 to 5 days prior to the second apheresis collection. The study day for N-803 administration will be determined based on the planned date of the second apheresis collection.
  Interventions: Drug: N-803

INTERVENTIONS:
Drug: N-803 — fixed dose of 1 mg by subcutaneous (SC) injection

SUMMARY:
This is phase 1 single cohort study evaluating the effects of N-803 administration on mononuclear cells (MNC) collected from healthy donors undergoing a procedure called apheresis.

DETAILED DESCRIPTION:
This phase 1, single cohort study will enroll up to 10 healthy subjects. All subjects will be pre-screened for eligibility. If the subject meets eligibility for study participation, informed consent will be obtained. Screening will include a history and physical, review of concomitant medications, assessment of NYHA functional status, assessment of ECOG performance status, clinical laboratory tests, pregnancy test (for women of child-bearing abilities), assessment of peripheral venous access, and a donor history questionnaire (DHQ). If subjects meet eligibility criteria, they will be asked to undergo two apheresis collections and donate their mononuclear cells (MNCs) for research purposes.

Subjects will be scheduled for the first apheresis collection on study Day 1. Two total blood volume (TBV) will be processed during each apheresis collections, which is currently the collection centers standard practice. All subjects will receive N-803 at a fixed dose of 1 mg by subcutaneous (SC) injection 4 to 5 days prior to the second apheresis collection. The N-803 dose may be administered starting on study Day 8 but no later than study Day 24. The study day for N-803 administration will be determined based on the planned date of the second apheresis collection. The second apheresis collection should occur between study Day 12 and study Day 29. Two TBV will be processed during this collection.

Subjects will be followed for collection of adverse events (AEs) from study Day 1 (first apheresis collection) through the end of study (EOS) visit. Subjects will be instructed to contact the study team in the event they experience AEs post N-803 administration (e.g., injection site reaction). In addition, AEs will be elicited from subjects during follow-up phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Healthy donors must be free of acute or chronic medical conditions (e.g., hypertension, kidney disease, diabetes, autoimmune disease, cardiovascular disease).
* Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
* Adequate organ function, evidenced by the following laboratory results:

Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3 Platelet count ≥ 100,000 cells/mm3 Hemoglobin ≥ 9.0 g/dL Total bilirubin ≤ 1.5 x upper limit of normal (ULN); unless the subject has documented Gilbert's syndrome Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 3 x ULN Serum creatinine ≤ 2.0 mg/dL or 177 μmol/L

* Adequate peripheral venous access.
* Must be able to be in the clinic for up to 6 hours on the day of collection.
* Must be able to sit or recline with limited movement for approximately 2-3 hours.
* Must agree to provide blood samples for clinical testing and immunological analysis.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0.

Exclusion Criteria:

* Received systemic antibiotics within 14 days prior to apheresis collection.
* New York Heart Association (NYHA) functional assessment score of > Class I.
* Any medical diagnosis that would prevent the donation of WBCs.
* History of or active human immunodeficiency virus (HIV).
* Active hepatitis B or hepatitis C.
* Have been advised by a medical provider not to donate blood.
* Women who are pregnant or breastfeeding. A negative serum pregnancy test in women of child-bearing potential is required at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAEs) and overall adverse events (AEs) coded in MedDRA | Study Day 1 through End of Study, assessed up to 45 days
  Incidence of SAEs and overall AEs coded in MedDRA

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAEs) and overall adverse events (AEs) graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (v5.0) | Study Day 1 through End of Study, assessed up to 45 days
  Incidence of SAEs and overall AEs graded using the NCI CTCAE v5.0
Evaluate and compare peripheral blood pre-apheresis and apheresis products collected without N-803 administration (unstimulated) and with N-803 administration (stimulated): - Percentage of NK cells | Study Day 1 through Study Day 24, assessed up to 24 days
  - Percentage of NK cells as measured by flow cytometry.
Evaluate and compare peripheral blood pre-apheresis and apheresis products collected without N-803 administration (unstimulated) and with N-803 administration (stimulated): - Immune profile | Study Day 1 through Study Day 24, assessed up to 24 days
  - Function and cell receptor profile of NK cells as measured by intracellular staining for cytokines, surface marker staining and assessments of cytotoxicity.
Evaluate and compare peripheral blood pre-apheresis and apheresis products collected without N-803 administration (unstimulated) and with N-803 administration (stimulated): - Serum cytokines | Study Day 1 through Study Day 24, assessed up to 24 days
  - Serum Cytokines

OTHER OUTCOMES:
Evaluate + compare the ex vivo expansion + enrichment of NK cells collected by apheresis without N-803 (unstimulated) + with N-803 administration (stimulated) via frequency, number, and phenotype of immune cells measured by flow + mass cytometry. | Study Day 1 through Study Day 24, assessed up to 24 days
  - Frequency, number, and phenotype of immune cells as measured by flow and mass cytometry.
Exploratory Objective: Evaluate and compare the ex vivo expansion and enrichment of NK cells collected by apheresis without N-803 (unstimulated) and with N-803 administration (stimulated) via Number of days to manufacture CENK and M-CENK. | Study Day 1 through Study Day 24, assessed up to 24 days
  - Number of days to manufacture CENK and M-CENK.
Exploratory Objective: Evaluate and compare the ex vivo expansion and enrichment of NK cells collected by apheresis without N-803 (unstimulated) and with N-803 administration (stimulated via Quality of CENK and M-CENK cells manufactured. | Study Day 1 through Study Day 24, assessed up to 24 days
  - Quality of CENK and M-CENK cells manufactured measured by the percentage of CD56 adequate for infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Sender, MD, Study Director — ImmunityBio, Inc.
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States